CLINICAL TRIAL: NCT06232031
Title: The Effect of Active Breathing Exercises on Swallowing Function for Elderly People in the Community: A Preliminary Self-control Study
Brief Title: The Effect of Active Breathing Exercises for Elderly People in the Community
Acronym: ABE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-KY-0120
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The observation group (Experimental): The observation group is the only group of the participants.The elderly individuals will be arranged to undergo a continuous three-week (21 days) duration of Active Breathing Exercises, with weekends off and training conducted only on weekdays. Apart from this,we require participants to only engage in daily activities and avoid strenuous and dangerous behaviors.
  Interventions: Behavioral: Active Breathing Exercises

INTERVENTIONS:
Behavioral: Active Breathing Exercises — Active breathing exercises aim to enhance the strength and flexibility of respiratory muscles through a series of exercises, improving breathing patterns and increasing respiratory efficiency. The following are common components of active breathing exercises: 1) Deep Breathing. 2) Chest Expansion. 3) Diaphragmatic Breathing. 4) Coughing Techniques. 5) Expiratory Resistance Training. 6) Gradual Increase in Activity.

SUMMARY:
The goal of this clinical trial is to explore the impact of Active Breathing Exercises on swallowing function and quality of life in community-dwelling elderly individuals (≥60 year old) with swallowing disorders. It primarily aims to address two key aspects: 1) the prevalence of dysphagia among community-dwelling elderly individuals, and 2) the effects of Active Breathing Exercises on swallowing function and quality of life in community-dwelling elderly individuals with swallowing disorders. All participants enrolled are required to undergo a continuous three-week (21 days) Active Breathing Exercises, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 15-30 minutes each.

DETAILED DESCRIPTION:
The investigators have designed a simple and user-friendly training method called "Active Breathing Exercises" based on commonly used swallowing training techniques in the department of rehabilitation medicine and the prevalent pathological causes of swallowing disorders in the elderly. The goal of this clinical trial is to explore the impact of Active Breathing Exercises on swallowing function and quality of life in community-dwelling elderly individuals (≥60 year old) with swallowing disorders. It primarily aims to address two key aspects: 1) the prevalence of dysphagia among community-dwelling elderly individuals, and 2) the effects of Active Breathing Exercises on swallowing function and quality of life in community-dwelling elderly individuals with swallowing disorders. All participants enrolled are required to undergo a continuous three-week (21 days) Active Breathing Exercises, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 15-30 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years old.
* No hospitalization within the past six months.
* With clear consciousness and able to cooperate with questionnaires and training.
* The elderly people who voluntarily participate and agree to adhere until the end of the study.

Exclusion Criteria:

* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Physical disability.
* Difficulty in mobility.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Eating Assessment Tool-10 | day 1 and day 21
  Eating Assessment Tool-10 is a scale used to evaluate swallowing function problems, and is one of the commonly used tools for assessing the swallowing ability of elderly individuals. Eating Assessment Tool-10 stands for 'Eating Assessment Tool-10', and was developed by professional medical institutions in the United States with the aim of quickly assessing potential difficulties and problems during the process of swallowing.The Eating Assessment Tool-10 scale consists of 10 questions that cover different aspects of swallowing function. Each question has a rating score ranging from 0 to 4, indicating the severity of difficulty in swallowing, with 0 representing no problem and 4 representing severe difficulty. The higher the total score, the more severe the swallowing function problem.

SECONDARY OUTCOMES:
Time consumed in eating | day 1 and day 21
  We require participants to eat a lunch according to their daily intake and habits, and count the time consumed
Water Swallow Test | day 1 and day 21
  The Water Swallow Test was recruited to assess swallowing function in participants at admission. Specifically, participants were instructed to sit and drink 30 ml of warm water. A 5-point scoring system is used as follows:
  1. Point: Successful swallowing of water within 5 seconds without coughing.
  2. Points: Able to swallow the water once but taking more than 5 seconds or swallowing in two or more attempts without coughing.
  3. Points: Able to swallow the water once with coughing.
  4. Points: Able to swallow the water in two or more attempts with coughing.
  5. Points: Unable to swallow all of the water, frequent coughing. The higher points indicate the worse swallowing function
Swallowing-Related Quality of Life Questionnaire | day 1 and day 21
  The Swallowing-Related Quality of Life Questionnaire (SWAL-QOL) is a validated tool used to assess the impact of swallowing difficulties on quality of life. It is a 44-item questionnaire designed to measure the physical, emotional, and social domains of swallowing-related quality of life.The higher final scores indicate the better life quality. The total score will be converted into a standard percentage

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group located in Miami

IPD SHARING:
Plan to Share IPD: No